CLINICAL TRIAL: NCT03182309
Title: The Prevalence, Disease Course, Prognosis and Interaction of Chronic Obstructive Pulmonary Disease With Sleep Apnea Hypopnea Syndrome
Brief Title: Registry for Chronic Obstructive Pulmonary Disease With Sleep Apnea Hypopnea Syndrome in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016YFC1304403
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: COPD; Sleep Apnea Syndromes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COPD and sleep apnea dyspnea syndrome represent two of the most common chronic lung diseases. It is reported that the prevalence of COPD with sleep apnea dyspnea syndrome is also very high. COPD and sleep apnea may have pathological or genetics interactions so that patients having both disorders tend to have worse outcomes than either condition alone. Data reflecting the prevalence, disease course and outcome of overlap syndrome is very limited in China. Therefore, the aim of the study is to describe the prevalence, treatment and outcome in Chinese patients and exploring the underlying interaction mechanism.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with informed consent

Exclusion Criteria:

* pregnant patients, patients with serious respiratory diseases other than COPD, patients with limited life expectancy, patients that can't coordinate well

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive COPD patients in 10 participating centers in China
Sampling Method: Non-Probability Sample
Enrollment: 3502 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD acute exacerbation | 3 years
  record the exacerbation events and related hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao Z, Zhang D, Sun H, Chang D, Lv X, Lin J, Liu J, Wu X, Hu K, Guo X, Tong Z. Anxiety and depression in patients with chronic obstructive pulmonary disease and obstructive sleep apnea: the overlap syndrome. Sleep Breath. 2022 Dec;26(4):1603-1611. doi: 10.1007/s11325-021-02500-2. Epub 2021 Nov 16. PMID 34783978
- [Derived] Zhu J, Zhao Z, Wu B, Shi Z, Nie Q, Fu Z, Zeng Z, Hu W, Dong M, Xiong M, Hu K. Effect of Body Mass Index on Lung Function in Chinese Patients with Chronic Obstructive Pulmonary Disease: A Multicenter Cross-Sectional Study. Int J Chron Obstruct Pulmon Dis. 2020 Oct 13;15:2477-2486. doi: 10.2147/COPD.S265676. eCollection 2020. PMID 33116464
- [Derived] Hu W, Dong M, Xiong M, Zhao D, Zhao Y, Wang M, Wang T, Liu Z, Lu L, Hu K. Clinical Courses and Outcomes of Patients with Chronic Obstructive Pulmonary Disease During the COVID-19 Epidemic in Hubei, China. Int J Chron Obstruct Pulmon Dis. 2020 Sep 23;15:2237-2248. doi: 10.2147/COPD.S265004. eCollection 2020. PMID 33061341
- [Derived] Zhu J, Zhao Z, Nie Q, Wang Y, Fu Z, Guo X, Hu K. Effect of lung function on the apnea-hypopnea index in patients with overlap syndrome: a multicenter cross-sectional study. Sleep Breath. 2020 Sep;24(3):1059-1066. doi: 10.1007/s11325-019-01961-w. Epub 2019 Nov 25. PMID 31768930